CLINICAL TRIAL: NCT03335683
Title: The Effects of a Phytotherapy Agent in Third Molar Surgery: a Split-mouth, Prospective, Randomized Study
Brief Title: Phytotherapy Agent in Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gaetano Isola, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Gaetano Isola, DDS, PhD, Dr. Gaetano Isola, University of Messina
Organization: University of Messina (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09/17
Record Dates: First submitted 2017-10-29; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Oral Soft Tissue Conditions
MeSH Terms: interventions — Lenidase

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phytoterapy agent (Experimental): Subjects were allocated to receive 1 h and 12 h after surgery: group 1, Lenidase® (Enfarma SRL, Misterbianco, Italy)
  Interventions: Drug: Lenidase
- Placebo (Placebo Comparator): Subjects were allocated to received 1 h and 12 h after surgery: placebo (Sugar pill, Sucratol - Placebo Capsules).
  Interventions: Drug: Lenidase

INTERVENTIONS:
Drug: Lenidase — drug per os twice day for 7 days, or for 10 days
  Other Names: Placebo

SUMMARY:
The aim of the present study was to evaluate the effect of a phytotherapy agent on clinical and inflammatory parameters, for the postoperative therapy of the impacted third molar surgery. The null hypothesis to invalidate was that, after the last follow-up, there were no variations between the phytotherapy agent and the placebo.

DETAILED DESCRIPTION:
The inclusion criteria were: (1) age between 18 and 32 years; (2) good general health; (3) the presence of two asymptomatic mandibular third molars with Class II position, type B impaction (Pell and Gregory, 1933), with similar root formation characteristics and position between the two sides; (4) absence of pericoronitis or signs of inflammation during the last 30 days. Orthopantomography (OPT) was used to determine tooth position. The exclusion criteria were (1) any systemic condition which might affect the study; (2) taking medications; (3) use of hormonal contraceptives; (4) medication by anti-inflammatory and immunosuppressive drugs; (5) status of pregnancy or lactation; (6) previous history of excessive drinking; (7) allergy to local anesthetic; (8) smoking.

The study was performed according to the CONSORT (Consolidated Standards Of Reporting Trials) guidelines. Patients who did not attend the second surgery or were unable to follow the study protocol were excluded, as were those whose surgical time exceeded 40 minutes.

Patients were scheduled for surgery in two separate clinical sessions (one side at a time), with a 1-month interval. Subjects were allocated to one of two groups according to the medication received 1 h and 12 h after surgery: group 1, Lenidase® (Enfarma SRL, Misterbianco, Italy); group 2, placebo (Sugar pill, Sucratol - Placebo Capsules). All patients in the study routinely received a prophylactic preoperative dose of oral antibiotic (1 g amoxicillin/clavulanic acid 1 hour before surgery) (Augmentin; GlaxoSmithKline, Verona, Italy).

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 30 years;
2. good general health;
3. the presence of two asymptomatic mandibular third molars with Class II position B impaction (Pell and Gregory, 1933), with similar root formation characteristics and position; absence of pericoronitis or signs of inflammation during the last 30 days. Ortopantomography (OPT) was used to determine tooth position.

Exclusion Criteria:

1. any systemic condition which might affect the study;
2. taking medications;
3. use of hormonal contraceptives;
4. medication by anti-inflammatory and immunosuppressive drugs;
5. status of pregnancy or lactation;
6. previous history of excessive drinking;
7. allergy to local anesthetic;
8. smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Pain | 10 days
  visual analogue scale (VAS), a score of 1 to 10. A score of 0 indicated no pain and 10, the worst pain.

SECONDARY OUTCOMES:
Swelling | 10 days
  Facial measure: swelling on the facial side receiving surgery. Measurement tragus to the nasal border (Tr-Al).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matarese, DDS, Study Director — Univeristy of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided